CLINICAL TRIAL: NCT05123950
Title: Treatment Patterns and Clinical Outcomes in First Line Recurrent/Metastatic Squamous Cell Carcinoma of the Head and Neck (1L R/M SCCHN) Patients in Europe
Brief Title: A Study of Treatment Patterns and Clinical Outcomes in First Line Recurrent/Metastatic Squamous Cell Carcinoma of the Head and Neck (1L R/M SCCHN) Participants in Europe
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-8HX
Record Dates: First submitted 2021-10-19; First posted 2021-11-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: Metastatic; Nivolumab; Recurrent; SCCHN; Treatment patterns; Outcomes
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Neoplasm Metastasis; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Participants diagnosed with R/M SCCHN between 01-Jan-2014 and 31-Dec-2016
- Cohort 1- Augment: Participants newly initiating 1L treatment for R/M SCCHN between 01-Jun-2017 and 01-Jun-2018

SUMMARY:
The purpose of this observational study is to collect real-world data that describes treatment patterns and clinical outcomes in participants with first line recurrent/metastatic squamous cell carcinoma of the head & neck (1L R/M SCCHN).

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

Participants are included in Cohort 1 - Augment if they meet the following criteria:

* Adults18 years or older
* Diagnosis of histologically confirmed R/M SCCHN, from any of the following primary sites only: oral cavity, oropharynx, hypopharynx, and larynx between 01-Jun-2017 and 31-June-2018.
* Prescribed 1L treatment for R/M SCCHN
* Treatment history and response available for medical chart abstraction from date of diagnosis until death or the end of the study in living participants
* Have available for review one month of follow-up data available post initiation of 1L R/M SCCHN therapy
* Informed consent form (ICF) signature/collection of living participants, as required by country regulation and local ethics committees

Participants are included in Cohort 1 if they meet the following criteria:

* Adults 18 years or older
* Diagnosis of histologically confirmed R/M SCCHN, from any of the following primary sites only: oral cavity, oropharynx, hypopharynx and larynx between 01-Jan-2014 and 31-Dec-2016.
* Prescribed 1L treatment for R/M SCCHN
* Treatment history and response available for medical chart abstraction from the date of diagnosis until death or the end of the study in living participants
* Have available for review one month of follow-up data post initiation of 1L R/M SCCHN therapy
* Informed consent form (ICF) signature/collection of living participants, as required by country regulation and local ethics committees

Exclusion Criteria:

Participants were excluded from either cohort if they meet the following criteria:

* Were enrolled in a cancer treatment-related clinical trial since the diagnosis of R/M SCCHN
* Recurrent or metastatic carcinoma of the nasopharynx, squamous cell carcinoma of unknown primary site, squamous cell carcinoma that originated from the skin and salivary gland or non-squamous histologies (e.g., mucosal melanoma).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A population of participants diagnosed with Recurrent/Metastatic Squamous cell carcinoma of the head and neck (R/M SCCHN) and treated with 1L therapy in two cohorts based on time period of initiating 1L treatment. Patients will be enrolled from France (FR), Germany (DE), and the United Kingdom (UK).
Sampling Method: Non-Probability Sample
Enrollment: 304 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-03-19 (Actual)

PRIMARY OUTCOMES:
Distribution of demographic characteristics of 1L R/M SCCHN participants treated with nivolumab: Age | At Baseline
  Recurrent/Metastatic (R/M) Squamous Cell Carcinoma of the Head & Neck (SCCHN)
Distribution of demographic characteristics of 1L R/M SCCHN participants treated with nivolumab: Height | At Baseline
Distribution of demographic characteristics of 1L R/M SCCHN participants treated with nivolumab: Weight | At Baseline
Distribution of demographic characteristics of 1L R/M SCCHN participants treated with nivolumab: Body surface area (BSA) | At Baseline
Distribution of demographic characteristics of 1L R/M SCCHN participants treated with nivolumab: Health insurance coverage | At Baseline
Distribution of demographic characteristics of 1L R/M SCCHN participants treated with nivolumab: Tobacco use | At Baseline
Distribution of demographic characteristics of 1L R/M SCCHN participants treated with nivolumab: Patient comorbidities | At Baseline
Distribution of demographic characteristics of 1L R/M SCCHN participants treated with nivolumab: Alcohol use | At Baseline
Distribution of clinical characteristics of 1L R/M SCCHN participants treated with nivolumab: Human papillomavirus(HPV) p -16 status | At Baseline
Distribution of clinical characteristics of 1L R/M SCCHN participants treated with nivolumab: Date of early stage diagnosis | At Baseline
Distribution of clinical characteristics of 1L R/M SCCHN participants treated with nivolumab: Receive a platinum-based agent for early stage diagnosis | At Baseline
Distribution of clinical characteristics of 1L R/M SCCHN participants treated with nivolumab: Receive radiation within 6 months prior to early stage diagnosis | At Baseline
Distribution of clinical characteristics of 1L R/M SCCHN participants treated with nivolumab: Undergo related surgeries within 6 months prior to early stage diagnosis | At Baseline
Distribution of clinical characteristics of 1L R/M SCCHN participants treated with nivolumab: Date of R/M SCCHN diagnosis | At Baseline
Distribution of clinical characteristics of 1L R/M SCCHN participants treated with nivolumab: Specialty of diagnosing physician | At Baseline
Distribution of clinical characteristics of 1L R/M SCCHN participants treated with nivolumab: Primary site of SCCHN at R/M diagnosis | At Baseline
Distribution of clinical characteristics of 1L R/M SCCHN participants treated with nivolumab: Clinical stage at R/M diagnosis | At Baseline
Distribution of clinical characteristics of 1L R/M SCCHN participants treated with nivolumab: Primary tumor stage at R/M diagnosis | At Baseline
Distribution of clinical characteristics of 1L R/M SCCHN participants treated with nivolumab: Lymph node involvement at R/M diagnosis | At Baseline
Distribution of clinical characteristics of 1L R/M SCCHN participants treated with nivolumab: Metastasis at R/M diagnosis | At Baseline
Distribution of clinical characteristics of 1L R/M SCCHN participants treated with nivolumab: Histologic tumor grade at R/M diagnosis | At Baseline
Distribution of clinical characteristics of 1L R/M SCCHN participants treated with nivolumab: Overall prognosis at R/M diagnosis | At Baseline
Distribution of clinical characteristics of 1L R/M SCCHN participants treated with nivolumab: Platinum-based grouping | At Baseline
Distribution of diagnostic procedures of 1L R/M SCCHN participants treated with nivolumab | At Baseline
Distribution of treatment patterns of 1L R/M SCCHN participants treated with nivolumab: First (second, third+) Line of therapy (LOT) | At Baseline
Distribution of treatment patterns of 1L R/M SCCHN participants treated with nivolumab: Duration of LOT | At Baseline
Distribution of treatment patterns of 1L R/M SCCHN participants treated with nivolumab: Administration form | At Baseline
Distribution of treatment patterns of 1L R/M SCCHN participants treated with nivolumab: Dose | At Baseline
Distribution of treatment patterns of 1L R/M SCCHN participants treated with nivolumab: Dose changes | At Baseline
Distribution of treatment patterns of 1L R/M SCCHN participants treated with nivolumab: Frequency of treatment regimen | At Baseline
Distribution of treatment patterns of 1L R/M SCCHN participants treated with nivolumab: Schedule of agent administration | At Baseline
Distribution of treatment patterns of 1L R/M SCCHN participants treated with nivolumab: Number of planned cycles | At Baseline
Distribution of treatment patterns of 1L R/M SCCHN participants treated with nivolumab: Number of completed cycles | At Baseline
Distribution of treatment patterns of 1L R/M SCCHN participants treated with nivolumab: Reasons for prescribing therapy | At Baseline
Distribution of treatment patterns of 1L R/M SCCHN participants treated with nivolumab: Reasons for discontinuing therapy | At Baseline
Distribution of treatment patterns of 1L R/M SCCHN participants treated with nivolumab: Dose delays | At Baseline
Distribution of treatment patterns of 1L R/M SCCHN participants treated with nivolumab: Radiation performed for R/M disease | At Baseline
Distribution of treatment patterns of 1L R/M SCCHN participants treated with nivolumab: Surgical procedures performed for R/M disease | At Baseline
Distribution of adverse events of 1L R/M SCCHN participants treated with nivolumab | At Baseline
Distribution of adverse events of 1L R/M SCCHN participants treated with nivolumab: Action taken | At Baseline
Distribution of adverse events of 1L R/M SCCHN participants treated with nivolumab: Resolution | At Baseline
Distribution of clinical outcomes of 1L R/M SCCHN participants treated with nivolumab: Response to therapy | At Baseline
Distribution of clinical outcomes of 1L R/M SCCHN participants treated with nivolumab: Duration of response | Up to approximately 36 months
Distribution of clinical outcomes of 1L R/M SCCHN participants treated with nivolumab: Overall survival | Up to approximately 36 months
Distribution of clinical outcomes of 1L R/M SCCHN participants treated with nivolumab: Progression free survival | Up to approximately 36 months

SECONDARY OUTCOMES:
Comparison of patient demographics, clinical characteristics, and treatment patterns between the Cohort 1- Augment and Cohort 1 | At Baseline
Comparison of time to event endpoints of OS, PFS, and DOR between Cohort 1- Augment and Cohort 1 | Up to approximately 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Medical Data Analytics, Parsippany, New Jersey, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm